CLINICAL TRIAL: NCT02277522
Title: Pilot Study of Redirected Autologous T Cells Engineered to Contain Anti-CD19 Linked to TCRζ and 4-1BB Signaling Domains in Patients With Chemotherapy Relapsed or Refractory Hodgkin Lymphoma
Brief Title: CD19 Redirected Autologous T Cells for Hodgkin Lymphoma
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: unable to meet enrollment goal
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 04414, 820840
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2017-11

CONDITIONS: Hodgkin Lymphoma With no Available Curative Treatment Options Who Have a Limited Prognosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RNA autologous T cells (anti CD19 CAR T cells) (Experimental)
  Interventions: Biological: RNA anti-CD19 CAR T cells

INTERVENTIONS:
Biological: RNA anti-CD19 CAR T cells — intravenously administered, RNA electroporated autologous T cells expressing CD19 chimeric antigen receptors expressing tandem TCRζ and 4-1BB (TCR /4-1BB) costimulatory domains (referred to as RNA CART19)

SUMMARY:
Pilot open-label study to estimate the feasibility, safety and efficacy of intravenously administered, RNA electroporated autologous T cells expressing CD19 chimeric antigen receptors expressing tandem TCR and 4-1BB (TCR /4-1BB) costimulatory domains (referred to as RNA CART19) in Hodgkin Lymphoma (HL) patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with HL with no available curative treatment options (such as autologous SCT) who have a limited prognosis (several months to < 2 year survival) with currently available therapies will be enrolled.

  i. HL with biopsy-proven relapse or refractory disease who are unresponsive to or intolerant of at least one line of standard salvage therapy ii. Patients must have evaluable disease by radiologic imaging (FDG PET/CT or PET/MRI) within 42 days of enrollment; evaluable includes both assessable and/or measurable disease as defined by Cheson et al., 2007.
* Age ≥ 18 years of age
* Creatinine < 1.6 mg/dl.
* ALT/AST < 3x upper limit of normal
* Bilirubin < 2.0 mg/dl, unless subject has Gilbert's syndrome (≤3.0 mg/dL)
* Patients with relapsed disease after prior allogeneic SCT (myeloablative or non-myeloablative) will be eligible if they meet all other inclusion criteria and

  1. Have no active GVHD and require no immunosuppression
  2. Are more than 6 months from transplant
* Performance status (ECOG) 0 or 1.
* Left Ventricular Ejection Fraction (LVEF) ≥ 40% as confirmed by ECHO/MUGA
* Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygen > 92% on room air
* Written informed consent is given.
* Successful T cell test expansion (to be performed as part of inclusion criteria until 3 subjects meet all enrollment criteria)

Exclusion Criteria:

* Pregnant or lactating women. The safety of this therapy on unborn children is not known. Female study participants of reproductive potential must have a negative serum pregnancy test at enrollment. A urine or serum pregnancy test will be performed within 72 hours before the first RNA CART19 infusion.
* Uncontrolled active infection.
* Active hepatitis B or hepatitis C infection.
* Any uncontrolled active medical disorder that would preclude participation as outlined.
* HIV infection.
* Patients with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system
* Patients with active CNS involvement by malignancy. Patients with prior CNS disease that has been effectively treated will be eligible providing treatment was >4 weeks before enrollment
* Patients in complete remission with no evidence of evaluable disease by radiologic imaging.
* History of allergy to murine proteins.
* History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40).
* Anti-CD20 monoclonal antibody therapy within the last 3 months, or absence of circulating B cells.
* Class III/IV cardiovascular disability according to the New York Heart Association Classification (see Appendix 1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-10; Primary Completion 2016-11 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Svoboda, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Svoboda J, Rheingold SR, Gill SI, Grupp SA, Lacey SF, Kulikovskaya I, Suhoski MM, Melenhorst JJ, Loudon B, Mato AR, Nasta SD, Landsburg DJ, Youngman MR, Levine BL, Porter DL, June CH, Schuster SJ. Nonviral RNA chimeric antigen receptor-modified T cells in patients with Hodgkin lymphoma. Blood. 2018 Sep 6;132(10):1022-1026. doi: 10.1182/blood-2018-03-837609. Epub 2018 Jun 20. PMID 29925499